CLINICAL TRIAL: NCT04446845
Title: Double vs. Single Stimulation in Young Poor Prognosis Patients Followed by a Fresh Embryo Transfer. A Randomized Clinical Trial
Brief Title: Double Stimulation Followed by a Fresh Embryo Transfer
Acronym: DUO_STIM_FRESH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundación Santiago Dexeus Font (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Organization: Fundacion Dexeus (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FSD-DUO-2020-02
Record Dates: First submitted 2020-06-19; First posted 2020-06-25 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — Follicular Phase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Double Stimulation (Elonva+rFSH) in luteal /follicular phase (Experimental): A first stimulation Stimulation will initiate in the luteal phase of the menstrual cycle On day 21 of the previous cycle150mcg of corifollitropin alfa (Elonva, Merck Sharp & Dohme (MSD), Spain) will be administrated and from day 8 of the stimulation when necessary, r-FSH of 250 IU per day will start until the day of ovulation trigger in a flexible gonadotropin-releasing hormone (GnRH) antagonist protocol. The first ovulation triggering will be induced with GnRH-agonist (triptorelin 0.2 ml). The embryos obtained from the first stimulation will be cryopreserved in a freeze-all approach.
  A second stimulation will start on day 2 of bleeding after the first oocyte retrieval.
  This time will correspond to a conventional COS where corifollitropin alfa will be administered on the beginning of the follicular phase, in a flexible antagonist protocol, and the second ovulation will be triggered with 250μg of Recombinant Human Chorionic Gonadotropin (rhCG)
  Interventions: Drug: Double Stimulation (Elonva+rFSH) in luteal /follicular phase
- Conventional Stimulation (Elonva+rFSH) in follicular phase (Active Comparator): A conventional COS where Corifollitropin alfa will be administered on the beginning of the follicular phase, in a flexible antagonist protocol, and the second ovulation will be triggered with 250μg of rhCG
  Interventions: Drug: Conventional Stimulation (Elonva+rFSH) in follicular phase

INTERVENTIONS:
Drug: Double Stimulation (Elonva+rFSH) in luteal /follicular phase — Following the 2nd oocyte retrieval, the patient will start luteal phase support (LPS) with vaginal micronized progesterone 200mg x 3 times a day until the day of the pregnancy test. All embryos will be cultured until day 5 in time-lapse incubators. In case of no blastocyst in the second cycle, or in case of poor embryo quality and in case of availability of frozen embryos from the first stimulation cycle, 1 frozen blastocyst from the first cycle will be thawed and will be transferred 5 days following the 2nd oocyte retrieval. Embryo transfer will be performed in all patients with available blastocysts, except in cases of high risk of ovarian hyperstimulation syndrome (OHSS) or progesterone elevation which is considered clinically relevant on the day of human chorionic gonadotropin (hCG) trigger, in which freeze-all strategy and deferred frozen embryo transferred will be considered.
  Arms: Double Stimulation (Elonva+rFSH) in luteal /follicular phase
Drug: Conventional Stimulation (Elonva+rFSH) in follicular phase — From the day of oocyte retrieval, the patients will be asked to start the LPS with vaginal micronized progesterone 3 times a day until the day of the pregnancy test. Embryo transfer will be performed in all patients with available blastocysts, except in cases of high risk of OHSS or progesterone elevation which is considered clinically relevant on the day of hCG trigger, in which freeze-all strategy and deferred frozen embryo transferred will be considered.
  Arms: Conventional Stimulation (Elonva+rFSH) in follicular phase

SUMMARY:
The major goal of controlled ovarian stimulation (COS) is to increase the number of oocytes harvested in order to result in the generation of a higher number of available embryos, extended embryo culture, embryo selection and finally providing higher cumulative live birth rates in infertile patients. Moreover, with the idea of the multiple waves of follicular production, we could start to take full advantage of the whole follicular cohort, and not only of the follicular wave.

In the context of low prognosis women such as women with poor ovarian response where, the success rates are very low due to the low number of oocytes retrieved and consequently of viable embryos), Dual stimulation may be of great value as a tool to improve outcomes.

The reported advantage of DuoStim is retrieved of more oocytes within a shorter time span, resulting in an increase in the probability of having transferable embryos increases, and theoretically reducing time to live birth as well as cycle cancellation.

DETAILED DESCRIPTION:
In assisted reproductive technologies (ART), despite the progress of the last decades, the achievement of a live birth still remains a challenge, especially for some categories of patients such as the one with poor ovarian reserve. One of the main tolls in reproductive medicine is controlled ovarian stimulation (COS) which is performed with the aim of obtaining multiple oocytes, so as to increase the chance of a live birth (LB) .

In order to induce multifollicular development in ovarian stimulation, recombinant FSH (or other products based on FSH) are given at the beginning of the follicular phase for an average of 10-12 days. The reason for this timing is mainly due to the fact that the follicular phase is clearly the moment when the ovaries are recruiting new follicles in order to establish the dominant for the cycle. However, as previously described follicular production by the ovaries follows a pattern of multicyclic waves. More specifically, a wave is a synchronous growth of follicles that have similar diameter and that can be documented with ultrasound . Beside the very well-known follicular wave (which is the one exploited in the COS), 64% of the women has two waves (follicular and luteal) and 32% of women has up to 3 waves in a normal cycle (early follicular, late follicular and luteal) .

The innovative concept of multiple waves of follicular development has been utilized in previous studies aiming to evaluate the effect of more than 1 stimulation cycles in a short period of time (less than 1 month). Specifically, two stimulation cycles have been performed in the same cycle by previous researcher (starting from the classical follicular COS and followed by a subsequent stimulation 5 days after the first oocyte retrieval) and it has been shown to be associated with improved cycle outcomes, alias higher number of oocytes retrieved and number of embryos obtained in total. Furthermore, in women with low ovarian response recent studies have suggested that the luteal phase stimulation appears to result in a higher number of oocytes retrieved as compared to the first follicular phase stimulation cycle .

Nevertheless, in spite of the accumulating evidence, a common characteristic of all of the published trials up to date is that in all of them dual stimulation cycle was initiated in the classical follicular phase followed by second stimulation cycle 5 days after oocytes retrieval. This approach had two major limitations:

1. Owing to this extended protocol and the luteal phase start the lack of synchronization between embryos and endometrium, a freeze-only protocol was considered essential to be adopted .
2. The fact that the 2nd stimulation cycle (luteal phase) always started 5 days after the first stimulation cycle does allow an unbiased evaluation of whether the improved outcomes on the second cycle are attributed to the luteal phase initiation of stimulation or to a carry-over effect of the first stimulation cycle.

Based on the above evidence we decided to design the current randomized trial which is, to our knowledge, the first to evaluate the benefit from the dual stimulation approach, not followed by a freeze-only strategy, but by fresh embryo transfer. In order to achieve this, we aim to compare the COS with the double stimulation (first luteal stimulation and then follicular ovarian stimulation) followed by fresh embryo transfer (ET) in poor prognosis patients undergoing in vitro fertilization/intra-cytoplasmatic sperm injections (IVF/ICSI) treatment.

The current randomized trial will allow us to

1. compare the double stimulation with a single stimulation strategy followed by fresh embryo transfer and
2. perform comparison of a luteal phase (1st cycle of the double stimulation group) and a follicular phase stimulation (control group) in a randomized setting

ELIGIBILITY:
Inclusion Criteria:

* Poor prognosis patients according to the POSEIDON group 3 & 4 (based on AMH)
* AMH <1.2
* age <40 years old
* BMI >18 and <35 kg/m2
* Body weight >50kg (in women <36 years old body weight >60kg)

Exclusion Criteria:

* Maternal age > 40 years
* History of untreated autoimmune, endocrine or metabolic disorders
* Previous ovarian cystectomy or oophorectomy
* Body weight <50kg (and body weight <60kg in women <36 years old)

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2020-10-30 (Actual); Primary Completion 2023-01-15 (Actual); Study Completion 2023-05-02 (Actual)

PRIMARY OUTCOMES:
Number of good-quality blastocysts | Day of embryo transfer (9 -20 days from initiation of the last ovarian stimulation)
  Embryo quality will be assessed according to the Istanbul consensus workshop criteria (Alpha Scientists in Reproductive Medicine and ESHRE Special Interest Human Reproduction 2011) and good quality embryo (GQE) at this developmental will be an expanded through to hatched blastocyst with an inner cell mass (ICM) that is prominent, easily discernible and consisting of many cells, with the cells compacted and tightly adhered together, and with a trophectoderm (TE) that comprises many cells forming a cohesive epithelium

SECONDARY OUTCOMES:
Number oocytes retrieved | 9 -20 days from initiation of the last ovarian stimulation
  The outcome will be evaluated on the day of oocyte retrieval
Number of cycles reaching the stage of embryo transfer | 9 -20 days from initiation of the last ovarian stimulation
  The outcome will be evaluated 5 days after last oocyte retrieval
Clinical pregnancy | 6-7 weeks of gestation
  The presence of intrauterine gestational sac with an embryonic pole demonstrating cardiac activity at 6-7 weeks of gestation
Ongoing pregnancy | 8-10 weeks of gestation
  The presence of intrauterine gestational sac with an embryonic pole demonstrating cardiac activity at 11-12 weeks of gestation
Time to pregnancy | 4-6 weeks of gestation
  Days between beginning of first stimulation and clinical pregnancy
Number of oocytes between follicular phase or luteal phase initiation of ovarian stimulation | 9 -20 days from initiation of the ovarian stimulation
  The outcome will be evaluated on the day of oocyte retrieval
Number of Metaphase II oocytes (MII) between follicular phase or luteal phase initiation of ovarian stimulation | 9 -20 days from initiation of the ovarian stimulation
  The outcome will be evaluated on the day of oocyte retrieval
Total additional dose of recombinant follicle stimulating hormone (rFSH) | 9 -20 days from initiation of the ovarian stimulation
  The outcome will be evaluated on the day of trigger
Length of stimulation | 9 -20 days from initiation of the ovarian stimulation
  The outcome will be evaluated on the day of trigger
Endocrine profile | Day 1, Day 6 , Day 8 of stimulation and Day of trigger 9 -20 days from initiation of the ovarian stimulation in each ovarian stimulation cycle
  Estradiol, Progesterone, luteinizing hormone (LH) and FSH

OTHER OUTCOMES:
Adverse events | Up to 30 days from treatment start date
  Any adverse event related with stimulation must be reported in Adverse Event Report Form

CONTACTS AND LOCATIONS:
Overall Officials: Nikolaos P Polyzos, MD PhD, Study Director — Hopital Universitari Dexeus
Locations (1):
- Hospital Universitario Quiron Dexeus, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alsbjerg B, Haahr T, Elbaek HO, Laursen R, Povlsen BB, Humaidan P. Dual stimulation using corifollitropin alfa in 54 Bologna criteria poor ovarian responders - a case series. Reprod Biomed Online. 2019 May;38(5):677-682. doi: 10.1016/j.rbmo.2019.01.007. Epub 2019 Jan 22. PMID 30795977
- [Background] Alpha Scientists in Reproductive Medicine and ESHRE Special Interest Group of Embryology. The Istanbul consensus workshop on embryo assessment: proceedings of an expert meeting. Hum Reprod. 2011 Jun;26(6):1270-83. doi: 10.1093/humrep/der037. Epub 2011 Apr 18. PMID 21502182
- [Background] Baerwald AR, Adams GP, Pierson RA. A new model for ovarian follicular development during the human menstrual cycle. Fertil Steril. 2003 Jul;80(1):116-22. doi: 10.1016/s0015-0282(03)00544-2. PMID 12849812
- [Background] Cardoso MCA, Evangelista A, Sartorio C, Vaz G, Werneck CLV, Guimaraes FM, Sa PG, Erthal MC. Can ovarian double-stimulation in the same menstrual cycle improve IVF outcomes? JBRA Assist Reprod. 2017 Sep 1;21(3):217-221. doi: 10.5935/1518-0557.20170042. PMID 28837031
- [Background] Coutifaris C. Freeze-only in vitro fertilization cycles for all? Fertil Steril. 2017 Aug;108(2):233-234. doi: 10.1016/j.fertnstert.2017.06.028. No abstract available. PMID 28778278
- [Background] Drakopoulos P, Blockeel C, Stoop D, Camus M, de Vos M, Tournaye H, Polyzos NP. Conventional ovarian stimulation and single embryo transfer for IVF/ICSI. How many oocytes do we need to maximize cumulative live birth rates after utilization of all fresh and frozen embryos? Hum Reprod. 2016 Feb;31(2):370-6. doi: 10.1093/humrep/dev316. Epub 2016 Jan 2. PMID 26724797
- [Background] Ferraretti AP, La Marca A, Fauser BC, Tarlatzis B, Nargund G, Gianaroli L; ESHRE working group on Poor Ovarian Response Definition. ESHRE consensus on the definition of 'poor response' to ovarian stimulation for in vitro fertilization: the Bologna criteria. Hum Reprod. 2011 Jul;26(7):1616-24. doi: 10.1093/humrep/der092. Epub 2011 Apr 19. PMID 21505041
- [Background] Kuang Y, Hong Q, Chen Q, Lyu Q, Ai A, Fu Y, Shoham Z. Luteal-phase ovarian stimulation is feasible for producing competent oocytes in women undergoing in vitro fertilization/intracytoplasmic sperm injection treatment, with optimal pregnancy outcomes in frozen-thawed embryo transfer cycles. Fertil Steril. 2014 Jan;101(1):105-11. doi: 10.1016/j.fertnstert.2013.09.007. Epub 2013 Oct 23. PMID 24161646
- [Background] Liu C, Jiang H, Zhang W, Yin H. Double ovarian stimulation during the follicular and luteal phase in women >/=38 years: a retrospective case-control study. Reprod Biomed Online. 2017 Dec;35(6):678-684. doi: 10.1016/j.rbmo.2017.08.019. Epub 2017 Aug 24. PMID 29030068
- [Background] Moffat R, Pirtea P, Gayet V, Wolf JP, Chapron C, de Ziegler D. Dual ovarian stimulation is a new viable option for enhancing the oocyte yield when the time for assisted reproductive technnology is limited. Reprod Biomed Online. 2014 Dec;29(6):659-61. doi: 10.1016/j.rbmo.2014.08.010. Epub 2014 Sep 4. PMID 25311972
- [Background] Morin SJ, Patounakis G, Juneau CR, Neal SA, Scott RT, Seli E. Diminished ovarian reserve and poor response to stimulation in patients <38 years old: a quantitative but not qualitative reduction in performance. Hum Reprod. 2018 Aug 1;33(8):1489-1498. doi: 10.1093/humrep/dey238. PMID 30010882
- [Background] Polyzos NP, Nwoye M, Corona R, Blockeel C, Stoop D, Haentjens P, Camus M, Tournaye H. Live birth rates in Bologna poor responders treated with ovarian stimulation for IVF/ICSI. Reprod Biomed Online. 2014 Apr;28(4):469-74. doi: 10.1016/j.rbmo.2013.11.010. Epub 2013 Dec 4. PMID 24581984
- [Background] Poseidon Group (Patient-Oriented Strategies Encompassing IndividualizeD Oocyte Number); Alviggi C, Andersen CY, Buehler K, Conforti A, De Placido G, Esteves SC, Fischer R, Galliano D, Polyzos NP, Sunkara SK, Ubaldi FM, Humaidan P. A new more detailed stratification of low responders to ovarian stimulation: from a poor ovarian response to a low prognosis concept. Fertil Steril. 2016 Jun;105(6):1452-3. doi: 10.1016/j.fertnstert.2016.02.005. Epub 2016 Feb 26. No abstract available. PMID 26921622
- [Background] Sighinolfi G, Sunkara SK, La Marca A. New strategies of ovarian stimulation based on the concept of ovarian follicular waves: From conventional to random and double stimulation. Reprod Biomed Online. 2018 Oct;37(4):489-497. doi: 10.1016/j.rbmo.2018.07.006. Epub 2018 Aug 11. PMID 30170909
- [Background] Tsampras N, Gould D, Fitzgerald CT. Double ovarian stimulation (DuoStim) protocol for fertility preservation in female oncology patients. Hum Fertil (Camb). 2017 Dec;20(4):248-253. doi: 10.1080/14647273.2017.1287433. Epub 2017 Feb 9. PMID 28423955
- [Background] Ubaldi FM, Capalbo A, Vaiarelli A, Cimadomo D, Colamaria S, Alviggi C, Trabucco E, Venturella R, Vajta G, Rienzi L. Follicular versus luteal phase ovarian stimulation during the same menstrual cycle (DuoStim) in a reduced ovarian reserve population results in a similar euploid blastocyst formation rate: new insight in ovarian reserve exploitation. Fertil Steril. 2016 Jun;105(6):1488-1495.e1. doi: 10.1016/j.fertnstert.2016.03.002. Epub 2016 Mar 25. PMID 27020168
- [Derived] Racca A, Rodriguez I, Garcia S, Arroyo G, Polyzos NP. Double versus single stimulation in young low prognosis patients followed by a fresh embryo transfer: a randomized controlled trial (DUOSTIM-fresh). Hum Reprod. 2024 Jun 6:deae104. doi: 10.1093/humrep/deae104. Online ahead of print. PMID 38845190
- See also: Related Info — http://dexeus.com